Optimization of the Bowel Preparation Regimen for Colon Capsule Endoscopy Procedure

Protocol ID: 2022-06303-02

Document date: 12/22/2022

# Information till forskningspersonerna

Vi vill fråga dig om du vill delta i ett forskningsprojekt. Innan du samtycker till att delta är det viktigt att du förstår varför undersökningen utförs och vad den innebär. Ta dig tid att noggrant läsa igenom nedanstående information. Diskutera den med undersökningspersonalen om det är något som är oklart. Diskutera gärna studien tillsammans med din familj eller husläkare om det känns tryggare.

I det här dokumentet får du information om projektet och vad det innebär att delta.

# Vad är det för projekt och varför vill ni att jag ska delta?

Mag- och tarmsjukdomar, såsom blödning, inflammation och tjocktarmstumörer, är vanligt förekommande och kan innebära betydande sjuklighet och även nedsatt livskvalitet. Kapselkoloskopi utvecklades för att diagnostisera mag- och tarmsjukdomar redan 2006 och har använts på vår mottagning sedan 2009.

Det är viktigt att tjocktarmen är tillräckligt rengjord för att full inspektion av tarmslemhinnan ska kunna göras. En fullständig kapselkoloskopi kräver att kapseln tar sig igenom hela mag-och tarmkanalen under kapselns batteritid (max 12 timmar). För detta krävs att tarmen är väl rengjord och att kapseln kan få hjälp att föras framåt genom tarmrörelsestimulerande medel.

Vår studie syftar till att undersöka och utvärdera effekten av ett förbättrat laxeringsprotokoll. Vår förhoppning är att den förbättrade laxeringsmetoden kommer att öka andelen kompletta undersökningar från tidigare 75% till 95%. Samtidigt förväntar vi oss att patienterna kommer att uppleva det mycket positivt att volymen laxermedel är mindre i det förbättrade laxeringsprotokollet.

Vi vill jämföra resultatet av tarmrengöring i redan utförda undersökningar där det tidigare protokollet användes med resultatet av undersökningar där det nu förbättrade protokollet för tarmrengöring används. Du har blivit remitterad för att genomgå en kapselundersökning och vid bedömningen av remissen ser vi att du uppfyller kriterierna för att kunna inkluderas i vår studie.

Projektet genomförs på Endoskopimottagningen på Skånes universitetssjukhus i Malmö. Forskningshuvudman för projektet är Region Skåne och ansvarig forskare är Ervin Toth (var god se nedan).

## Hur går studien till?

Du kommer att genomgå en kapselkoloskopi-undersökning enligt klinikens vanliga rutiner. Vi kommer att använda PillCam® kapselsystem, vilket är det system som används i vår rutinmässiga verksamhet. Det består av en liten videokapsel (11x31 mm), som innehåller två små kameror för bildtagning.

Du sväljer denna engångskapsel med ett glas vatten och den kommer direkt att börja ta bilder från mag-och tarmkanalen och överföra dem trådlöst, genom radiovågor till en inspelningsenhet, som du bär runt midjan. Kapseln tar sig sedan genom mag- och tarmkanalen med hjälp av tarmens normala rörelser och lämnar sedan kroppen via ändtarmen inom 6–12 timmar. De inspelade videofilmen kodas och bedöms i efterhand av läkaren, som då kan ställa en diagnos och fatta beslut om lämplig behandling.

Undersökningen innebär att tarmen först måste rengöras. Det sker med hjälp av att du dricker laxeringsmedlet Plenvu (0,5 liter) samt vatten (1 liter) på kvällen före undersökningsdagen och på morgonen på undersökningsdagen.

Under undersökningsdagen kvarstannar du på Endoskopimottagningen och dricker enligt protokollet två olika medel samt får mediciner vid behov för att föra kapseln snabbare genom mag- och tarmkanalen. Samtliga läkemedel som ingår i studien är sedan tidigare godkända och används i rutinmässig klinisk praktik.

Du kan hela tiden under kapselundersökningen vara uppegående och röra dig som vanligt. Du får hjälp och instruktioner av en endoskopisköterska under hela undersökningen. Det är viktigt att du under hela undersökningen talar om för oss om du känner av något ovanligt i ditt hälsotillstånd.

## Möjliga följder och risker med att delta i studien

Frånsett att du kommer att få inta en lägre volym laxermedel än vi vanligen ordinerar patienten vid kapselkoloskopi finns det ingen särskild fördel för dig som patient att delta i studien – mer än att du på detta sätt bidrar till forskningen inom mag- och tarmsjukdomar och optimeringen kapselundersökningar. Det finns samtidigt inga ökade risker för dig som patient att delta i studien, eftersom du oavsett är planerad att genomgå en kapselundersökning.

Som alltid vid kapselundersökningar finns en liten risk, som uppskattas till mindre än 1 procent, att kapseln inte kommer att komma ut med avföringen som förväntat. Detta kan inträffa om du har ett trängre parti i matsmältningssystemet, som inte var känt innan undersökningen. Ett sådant trängre område kan vi normalt misstänka finnas vid en känd sjukdom i mag- och tarmkanalen eller om patienten har genomgått någon form av kirurgiskt ingrepp i mag- och tarmkanalen. Om kapseln inte lämnar kroppen på normalt sätt och orsakar en blockering i mag- och tarmkanalen kan du drabbas av magsmärtor, illamående och kräkningar. Om kapseln inte kommer ut kan du behöva genomgå medicinsk behandling, endoskopisk undersökning eller kirurgi för att ta bort den. Detta är mycket ovanligt, men det är viktigt att du känner till att risken finns.

Eftersom du är remitterad till Endoskopimottagningen för att genomgå en kapselundersökning kommer vi att ha tillgång till din patientjournal, såsom är brukligt inom sjukvården. Dina journal- och personuppgifter hanteras enligt precis samma sekretessregler som vid ett vanligt sjukvårdsbesök. De uppgifterna, t ex ålder och kön, som vi använder i studien kommer aldrig kunna härröras specifikt till just dig utan uppgifterna används endast i studien på så kallad gruppnivå (t ex en viss åldersgrupp). Alla uppgifter från de personer som ingår i studien hanteras enligt gällande sekretessregler och förvaras säkert. Ingen obehörig kommer att få ta del av personuppgifter. Uppgifterna kommer att sparas minst 10 år efter publicering.

# Vad händer med mina uppgifter?

Projektet kommer att samla in och registrera information om dig. Denna information består dels av bakgrundsinformation om dig – såsom ålder och kön och relevanta tidigare diagnoser (t ex känd magoch tarmsjukdom) och dels bilderna från kapselundersökningen. Om du vill delta i denna studie innebär din underskrift att din medicinska information direkt kan göras åtkomlig för och granskas av behöriga personer som arbetar med studien eller representanter från tillsynsmyndigheter eller av den etiska kommittén. Syftet med inspektionen av denna registrering är att säkerställa att den information som insamlas under forskningsstudien är korrekt och att studiens protokoll har

genomförts på rätt sätt. Information som avslöjar din identitet kommer dock att hållas konfidentiell, utom i sällsynta undantagsfall då avslöjandet av din identitet till tredje part kan vara påkallad enligt lag eller i en rättsprocess. Information från studien kan komma att publiceras, men ditt namn kommer inte att tas med och dina uppgifter kommer inte att kunna härledas till dig.

Hanteringen av dina uppgifter regleras enligt dataskyddsförordningen för behandling av persondata (GDPR, General Data Protection Regulation), som började gälla den 25 maj 2018 i Sverige. Dina uppgifter är sekretesskyddade och ingen obehörig har tillgång till registret. Vid databearbetningen kommer namn och personnummer att ersättas med en kod så att du endast kan identifieras av den studieansvarige läkaren. Dina svar och dina resultat kommer att behandlas och sparas så att ingen obehörig kan ta del av dem.

Ansvarig för dina personuppgifter är Region Skåne. Enligt EU:s dataskyddsförordning har du rätt att kostnadsfritt få ta del av de uppgifter om dig som hanteras i studien, och vid behov få eventuella fel rättade. Du kan också begära att uppgifter om dig raderas samt att behandlingen av dina personuppgifter begränsas. Rätten till radering och till begränsning av behandling av personuppgifter gäller dock inte när uppgifterna är nödvändiga för den aktuella forskningen. Om du vill ta del av uppgifterna ska du kontakta huvudansvarig forskare (se nedan). Dataskyddsombud nås på 044-309 30 00 (Region Skåne, 291 89 Kristianstad, region@skane.se). Om du är missnöjd med hur dina personuppgifter behandlas har du rätt att inkomma med klagomål till Integritetsskyddsmyndigheten.

# Vad händer med mina prover?

Inga prover kommer att tas i den här studien.

#### Hur får jag information om resultatet av studien?

Resultaten från studien kommer att publiceras i internationella tidskrifter och presenteras vid kongresser. Om du vill kan du kontakta huvudansvarig forskare Ervin Toth (se nedan) för att erhålla en kopia på den publicerade artikeln. Önskar du även ta del av din individuella data är du också välkommen att kontakta ansvariga forskare (se nedan). Du har ingen skyldighet att behöva ta del av studiens resultat.

Om kapselundersökningen leder till eventuella oförutsedda fynd kommer du som patient att handläggas inom sjukvården enligt sedvanliga rutiner.

#### Försäkring och ersättning

Patientförsäkringen gäller för alla deltagarna i studien. Patientförsäkringen är en skattepliktig inkomst. Ingen ersättning kommer att betalas ut för deltagande i studien.

## Deltagandet är frivilligt

Ditt deltagande är frivilligt och du kan när som helst välja att avbryta deltagandet. Om du väljer att inte delta eller vill avbryta ditt deltagande behöver du inte uppge varför, och det kommer inte heller att påverka din framtida vård eller behandling.

# Utvärdering av ett optimerat tarmrengöringsprotokoll för kapselkoloskopi: en jämförande studie

Om du vill avbryta ditt deltagande ska du kontakta den ansvariga forskaren för studien (se nedan).

# Ansvarig forskare för studien

**Ervin Toth** 

Docent, överläkare

Skånes universitetssjukhus

Telefon: 072-587 78 82

E-post: <a href="mailto:ervin.toth@med.lu.se">ervin.toth@med.lu.se</a>

# Utvärdering av ett optimerat tarmrengöringsprotokoll för kapselkoloskopi: en jämförande studie

# Samtycke till att delta i studien Jag har fått muntlig och skriftlig information om studien och har haft möjlighet att ställa frågor. Jag får behålla den skriftliga informationen. Jag samtycker till att delta i studien Utvärdering av ett optimerat tarmrengöringsprotokoll för kapselkoloskopi: en jämförande studie. Jag samtycker till att uppgifter om mig behandlas på det sätt som beskrivs i forskningspersonsinformationen.

Underskrift

Plats och datum